CLINICAL TRIAL: NCT06260605
Title: The Effect of Diabetes Complications Education Given With Puzzles on the Knowledge Level of Nursing Students
Brief Title: Complications of Diabetes With Puzzles
Acronym: Diabetes with
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bilecik Seyh Edebali Universitesi (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Burcu Bayrak 1; Burcu (Registry Identifier: Bayrak)
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2023-12

CONDITIONS: Diabetes Complications
Keywords: nursing students; puzzles; diabetes
MeSH Terms: conditions — Diabetes Complications; Diabetes Mellitus | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nursing students (Experimental): Nursing students' education
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — Nursing students learning about diabetes complications

SUMMARY:
In this study, it was aimed to investigate the effect of diabetes complications training on endocrine system diseases and nursing care in the Internal Medicine Nursing course on the knowledge level of nursing students.

DETAILED DESCRIPTION:
Puzzles, which are among the active learning tools, are frequently preferred today because they make learning fun, are economical, improve problem-solving skills and offer understandable learning. The student's involvement in a fun game, his effort to find the correct information, and the feedback he receives afterwards have an important place in terms of learning. It develops students' decision-making power with a critical perspective. Puzzles increase students' motivation and self-confidence by turning complex concepts into a hobby. The use of the puzzle technique in learning concepts related to theoretical knowledge is among the studies carried out in recent years. The puzzle technique is used in many fields such as pharmacology in nursing education (Shawahna & Jaber, 2020), child health and diseases (Kaynak et al., 2023), pain management (Köse Tosunöz & Deniz Doğan, 2023), teaching in nursing (Kalkan et al., 2022). It has been shown to have a positive effect on learning information. In this study, it was aimed to investigate the effect of diabetes complications training on endocrine system diseases and nursing care in the Internal Medicine Nursing course on the knowledge level of nursing students.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in research
* Having course continuity

Exclusion Criteria:

* Not volunteering to participate in the research

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2023-12-19 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-03-04 (Actual)

PRIMARY OUTCOMES:
Education | 5 weeks
  Nursing students learning about diabetes complications

CONTACTS AND LOCATIONS:
Locations (1):
- Bilecik Şeyh Edebali University, Bilecik, Merkez, Turkey (Türkiye)